CLINICAL TRIAL: NCT01489033
Title: Multicentre Phase I Randomized Double Blind Placebo Controlled Study of Subcutaneous Immunotherapy in Subjects With Allergic Rhinoconjunctivitis ± Asthma Sensitised to Phleum Pratense.
Brief Title: Subcutaneous Immunotherapy in Patients Sensitized to Phleum Pratense
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roxall Medicina España S.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-PHL-P1-001; 2009-015000-26 (EudraCT Number)
Record Dates: First submitted 2011-12-07; First posted 2011-12-09 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Allergic Rhinoconjunctivitis
Keywords: Allergic rhinitis; Phleum pratense; Timothy grass pollen allergy; subcutaneous immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group A active (Experimental): 6 administrations and 5 weeks duration
  1. Vial 2: 0.1 ml, 0.2 ml and 0.5 ml at 1 week intervals
  2. Vial 3: 0.1 ml, 0.2 ml and 0.5 ml at 1 week intervals.
  Interventions: Biological: Subcutaneous immunotherapy with Phleum pratense pollen extract
- Group A placebo (Placebo Comparator): 6 administrations and 5 weeks duration
  1. Vial 2: 0.1 ml, 0.2 ml and 0.5 ml at 1 week intervals
  2. Vial 3: 0.1 ml, 0.2 ml and 0.5 ml at 1 week intervals.
  Interventions: Biological: Subcutaneous immunotherapy with Phleum pratense pollen extract
- Group B active (Experimental): 8 administrations and 7 weeks duration
  1. Vial 1: 0.2 ml at 1 week intervals
  2. Vial 2: 0.1 ml, 0.2 ml, 0.4 ml at 1 week intervals
  3. Vial 3: 0.1 ml, 0.2 ml, 0.4 ml and 0.5 ml at 1 week intervals
  Interventions: Biological: Subcutaneous immunotherapy with Phleum pratense pollen extract
- Group B placebo (Placebo Comparator): 8 administrations and 7 weeks duration
  1. Vial 1: 0.2 ml at 1 week intervals
  2. Vial 2: 0.1 ml, 0.2 ml, 0.4 ml at 1 week intervals
  3. Vial 3: 0.1 ml, 0.2 ml, 0.4 ml and 0.5 ml at 1 week intervals
  Interventions: Biological: Subcutaneous immunotherapy with Phleum pratense pollen extract
- Group C active (Experimental): 8 administrations, 2 administrations in the same day. 1 week interval between 2 doses, during 3 weeks.
  1. Week 1: vial 2 - 2 administrations of 0.1 ml with 30 minute interval
  2. Week 2: vial 2 - 0.2 ml and 0.3 ml with 30 minute interval
  3. Week 3: vial 3 - 2 dose of 0.1 ml with 30 minute interval
  4. Week 4: vial 3 - 0.2 ml and 0.3 ml with 30 minute interval
  Interventions: Biological: Subcutaneous immunotherapy with Phleum pratense pollen extract
- Group C placebo (Placebo Comparator): 8 administrations, 2 administrations in the same day. 1 week interval between 2 doses, during 3 weeks.
  1. Week 1: vial 2 - 2 administrations of 0.1 ml with 30 minute interval
  2. Week 2: vial 2 - 0.2 ml and 0.3 ml with 30 minute interval
  3. Week 3: vial 3 - 2 dose of 0.1 ml with 30 minute interval
  4. Week 4: vial 3 - 0.2 ml and 0.3 ml with 30 minute interval
  Interventions: Biological: Subcutaneous immunotherapy with Phleum pratense pollen extract

INTERVENTIONS:
Biological: Subcutaneous immunotherapy with Phleum pratense pollen extract — Increasing doses up to a maximum dose of 500 TSU

SUMMARY:
Based on EMA (European Medicines Agency) new guidelines on the clinical development of products for immunotherapy for the treatment of allergic disease the aim of this study was to assess safety and tolerability of three different subcutaneous immunotherapy dose escalations in patients allergic to the pollen of Phleum pratense.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must sign the informed consent form.
2. Patients must be between 18 and 60 years of age.
3. Patients who obtained a prick test result greater or equal to 3 mm diameter and a specific IgE greater or equal to class 2 (CAP/PHADIA) to Phleum pratense.
4. Patients with seasonal allergic rhinoconjunctivitis against Phleum pratense during a minimum of 2 years prior to study participation. Although allergic rhinoconjunctivitis is the pathology under study, the inclusion of patients with mild or moderate concomitant asthma is allowed.
5. Patients will preferably be monosensitized to Phleum pratense. Polysensitized patients to other seasonal allergens will be accepted if sensitizations are caused by Pollens whose seasons do not overlap with Phleum pratense.

   Polysensitized patients to perennial allergens will also be accepted if not clinically relevant during the study period.
6. Women of childbearing potential must have a negative urine pregnancy test at Screening visit/Visit 0
7. Women of childbearing potential must agree to use an appropriate contraception method during the study if they are sexually active.

Exclusion Criteria:

1. Stable and continued use of medication for allergic pathology during 2 weeks prior to inclusion.
2. Patients sensitised to other overlapping seasonal allergens and with specific IgE levels greater or equal to class 2 CAP/PHADIA.
3. Patients who received immunotherapy in the previous 5 years for Phleum pratense or for any allergen with cross reactivity or patients that are currently receiving immunotherapy for any allergen.
4. Patients with severe asthma or FEV1 lower than 60% or asthma requiring inhaled or systemic corticoid treatment at the time of study entry or within 8 weeks prior to treatment commencement.
5. Patients with: immunological, cardiac, renal or hepatic illnesses or any other medical condition that the investigator deems relevant so as to interfere with the study.
6. Patients with a previous history of anaphylaxis
7. Patients with unstable angina
8. Patients with uncontrolled hypertension
9. Patients with clinically significant arrythmias
10. Patients with neoplasia
11. Patients with clinically relevant malformations of the upper respiratory tract.
12. Other chronic or immunological disease that could interfere with the assessment of the investigation product or that could generate any additional risk for the patient
13. Patients who have participated in another clinical trial within 3 month prior to enrolment.
14. Patients under treatment with tricyclic antidepressives, psychotropics or beta-blockers
15. Female patients who are pregnant or breast-feeding or women of childbearing potential that do not agree to use an appropriate contraception method during the study if they are sexually active, if they have not been surgical sterilised or present any other incapacity to bear
16. Patient who does not attend the visits
17. Patient's lack of collaboration or refusal to participate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Number and seriousness of both local and systemic adverse reactions | From informed consent signature (V0) until the end of patient participation in the study (depending on the treatment assigned between 4 and 8 weeks )

SECONDARY OUTCOMES:
Immunoglobulin levels (IgE specific, IgG total and IgG4) and prick test dose response | Before (V0) and after treatment (depending on the treatment assigned between 4 and 8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Álvarez-Cuesta, Md, PhD, Principal Investigator — Hospital Universitario Ramon y Cajal
Locations (1):
- Hospital Ramón y Cajal, Madrid, Spain